CLINICAL TRIAL: NCT00445276
Title: Efficacy Study of Diacerein in the Symptomatic Treatment of Knee Osteoarthritis
Brief Title: Symptomatic Efficacy of Diacerein in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires NEGMA (Industry)
Responsible Party: Patrick Darses, Negam-Lerads
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEC / ART 05 566 N; AFSSAPS:050984; CCPPRB:2005-27
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Diacerein; Painful osteoarthritis; Clinical trial
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — diacerein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Diacerein

SUMMARY:
Pain is the main symptom of osteoarthritis that motivates medical visits. Diacerhein has already demonstrated its efficacy in knee and/or hip osteoarthritis. This study aims at confirming the efficacy of diacerhein in symptomatic knee osteoarthritis using known and validated criteria and according to the recommendations and guidelines for this kind of study.

ELIGIBILITY:
Inclusion Criteria:

* Painful primary osteoarthritis (VAS ≥ 40 mm)
* Radiologically proven (Kellgren & Lawrence grade I to III)
* Requiring the prescription of a symptomatic treatment of pain

Exclusion Criteria:

* Severe associated diseases
* Wash-out: AINS, Coxibs, Paracetamol, anti-osteoarthritic treatments, hyaluronic acid, knee tidal lavage
* Other osteoarticular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
VAS on pain movement, WOMAC A 1.1 section

SECONDARY OUTCOMES:
WOMAC : total, pain, physical function
Paracetamol consumption
Global assessment of the patient
Responder patients with OMERACT-OARSI criteria
Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Jean - Pierre Valat, Principal Investigator — Unafilliated
Locations (1):
- Chu Trousseau, Tours, France